CLINICAL TRIAL: NCT02963181
Title: Identifying the Pathophysiology of Neurogenic Orthostatic Hypotension and the Effects of Melatonin on Reducing Supine Hypertension in Peripherally Intact Versus Denervated Post-ganglionic Sympathetic Nerves
Brief Title: Effects of Melatonin to Reduce Nocturnal Hypertension in Patients With Neurogenic Orthostatic Hypotension
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI leaving
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 010788
Record Dates: First submitted 2016-11-07; First posted 2016-11-15 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2018-03

CONDITIONS: Hypotension, Orthostatic; Hypertension; Autonomic Nervous System Diseases
Keywords: Melatonin; Yohimbine; Anti-hypertensive agents
MeSH Terms: conditions — Hypotension, Orthostatic; Hypertension; Autonomic Nervous System Diseases | interventions — Yohimbine; Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effects of Yohimbine (Experimental): Investigation into the integrity of post-ganglionic sympathetic nerves in patients with idiopathic neurogenic orthostatic hypotension
  Interventions: Drug: Yohimbine
- Effects of melatonin on blood pressure (Experimental): Investigation into the effects of melatonin at two separate dosages (2 and 5mg) on nocturnal blood pressure in NOH patients with intact versus denervated post-ganglionic sympathetic nerves
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Yohimbine — Oral Yohimbine will be used to identify the integrity of post-ganglionic sympathetic nerves in patients with NOH
  Other Names: DIN:01901885
  Arms: Effects of Yohimbine
Drug: Melatonin — Monitor the effects of melatonin on supine hypertension in NOH patients with intact and denervated post-ganglionic nerves.
  Identify the mechanistic pathway of melatonin in blood pressure regulation
  Other Names: melatonin timed release; 2 or 5 mg
  Arms: Effects of melatonin on blood pressure

SUMMARY:
Neurogenic Orthostatic Hypotension (NOH) is clinically defined as a consistent drop in systolic blood pressure (SBP) ≥30mmHg upon standing from a seated or lying position. However, 50% of NOH patients also have associated supine hypertension. It has been proposed that supine hypertension is the result of intact post-ganglionic sympathetic nerves and therefore due to residual sympathetic tone. Furthermore, research investigating the effects of melatonin shows blood pressure implication of this naturally secreted hormone. Specifically, melatonin has been investigated as a non-traditional anti-hypertensive agent for patients with essential and nocturnal hypertension. Central and peripheral mechanisms have been proposed to help explain how melatonin reduces blood pressures. Therefore, we aim to identify NOH patients as having either intact or denervated post-ganglionic sympathetic nerves, monitor the correlation to supine hypertension and subsequently investigate the effects of melatonin on blood pressure in these patients.

DETAILED DESCRIPTION:
Neurogenic orthostatic hypotension (NOH) is a debilitating condition associated with reduced quality of life, impaired function and is also an independent predictor of mortality(Bendini et al., 2007; Cordeiro et al., 2009; Rose et al., 2006). NOH is clinically defined as a sustained reduction in systolic blood pressure (SBP) ≥30mmHg within 3 minutes of standing or head-up tilt to at least 60 degrees on a tilt table(Freeman et al., 2011). Specifically, neurogenic OH can be differentiated from other causes of orthostatic hypotension, such as hypotension due to endocrine issues, generalized low blood pressure, low blood volume, etc., in that NOH is associated with autonomic dysfunction. Specifically, dysfunction of the reflexive regulation mediated by the sympathetic nervous system(Goldstein and Sharabi, 2009; Low et al., 2008).

Studies have implicated specific dysfunction of the peripheral sympathetic nerves in disorders that have accompanying NOH such as Multiple System Atrophy (MSA), Pure Autonomic Failure (PAF) and Parkinson Disease (PD+NOH)(Imrich et al., 2009; Senard et al., 1993; Sharabi et al., 2006). In clinical NOH populations with known diagnoses such as MSA, PAF and PD+NOH, infusions of yohimbine have been used to detect whether post-ganglionic sympathetic nerves are intact or denervated. Yohimbine is an alpha-adrenoceptor antagonist that, in healthy/intact sympathetic nerves, causes an increase in the release of norepinephrine (NE) from sympathetic nerves via increased sympathetic neuronal outflow. NE is a natural neurotransmitter that is released when the sympathetic nervous system is required to increase its activity. In persons with intact post-ganglionic sympathetic nerves an infusion of yohimbine results in an increase in blood pressure, arterial NE levels, and heart rate levels, with a decrease in forearm blood flow indicative of vasoconstriction. In contrast, patients with sympathetic denervation these responses are attenuated(Senard et al., 1993; Shannon et al., 2000; Sharabi et al., 2006). However, in these studies, the clinical population consisted of MSA, PAF and PD+NOH. Little research has been done in NOH populations without an underlying diagnosis, and in fact, 1/3 of patients with NOH have no identifiable underlying cause (Robertson and Robertson, 1994).

Furthermore, it has been hypothesized that supine hypertension in this select patient population is due to residual sympathetic tone in patients with intact post-ganglionic sympathetic nerves. Approximately 50% of NOH patients have associated supine hypertension(Shannon et al., 2000), which if left untreated, comes with its very own unique set of cardiovascular complications, such as significantly higher left-ventricular mass indices, specific end organ damage(Vagaonescu et al., 2000), heart attack and stroke. Therefore, clinicians are left with the challenging dilemma of finding a near impossible balance between the risks associated with supine hypertension versus the risks of sudden hypotension upon standing and the associated consequences of falls, fractures and head injuries resulting in more immediately morbid events. Medications such as nitrates and other antihypertensives can be prescribed, however their use is strongly cautioned as it is quite frequent that NOH patients are often older and have nocturia, and as a result are up frequently throughout the night. Other options such as raising the head of the bed 4 inches from the ground in order to reduced renal hyper-perfusion pose as an additional conservative measure, however, this does not act as a treatment for the supine hypertension.

In contrast, melatonin is a natural hormone secreted by the pineal gland in response to low light and is involved in maintaining proper circadian rhythms and sleep patterns. However, more recently, there has been a growing source of literature supporting melatonin as having an important role in blood pressure control: i) In rats, following pinealectomy, there is evidence of vasoconstriction (Cunnane et al., 1980) and hypertension (Zanoboni et al., 1978; Zanoboni and Zanoboni-Muciaccia, 1967). ii) Experimental hypertension elicited via pinealectomy can be reversed through exogenous administration of melatonin(Holmes and Sugden, 1976). iii) Continuous light exposure, results in a melatonin deficiency, peripheral vasoconstriction and hypertension(Briaud et al., 2004; Brown et al., 1991).

Therefore, melatonin is now being looked at as a non-traditional anti-hypertensive medication in patients with essential and nocturnal hypertension. In a study of 34 patients with nocturnal hypertension, administration of melatonin proved to have a slight, yet significant, reduction in nighttime blood pressure measurements(Grossman et al., 2006). In these studies, melatonin was taken for 3 or 4 weeks via an oral prescription 1 hour before bed. The dose was formulated as a controlled- or slow-release throughout the night. In these studies, there was an average systolic BP drop of 6.5mmHg and 4mmHg diastolic in supine/nighttime blood pressures. While this reduction may not seem significant, clinical it is. In a study of 2156 hypertensive patients, following a median follow-up period of 5.6 years it was found that the cardiovascular risk adjustment per 5mmHg reduction of nocturnal blood pressure in patients aged 55 years and above, was 0.92 (95%CI0.88-0.96) and per 5mmHg reduction in nocturnal diastolic blood pressure was 0.82 (95%CI0.77-0.88). The decrease in mean asleep BP during follow-up was most significantly associated with event-free survival (Hermida et al., 2010). In women, a mean decrease of 6mmHg in diastolic pressure significantly reduced overall mortality from vascular disease by 21%, fatal and nonfatal stroke by 42%, and fatal and nonfatal coronary heart disease by 14% (Rich-Ewards et al., 1995). Currently, the posed mechanisms of melatonin to reduced blood pressure consist of both central and peripheral mechanisms (Capsoni et al., 1994; Pogan et al., 2002; Ray, 2003; Satake et al., 1991; Stankov et al., 1993; Weekley, 1993). Therefore, the objectives of the current study are: 1. Identify NOH patients as having either peripherally intact vs denervated post-ganglionic sympathetic innervation to help identify a group of patients potentially more susceptible to supine hypertension. 2. Administer melatonin and monitor its effects on supine/nocturnal blood pressures in patients with supine hypertension, and 3. Investigate the proposed mechanisms of melatonin by comparing its effects in patients with peripherally intact vs denervated sympathetic nerves.

ELIGIBILITY:
Inclusion Criteria:

* Control population: Healthy males or females between the ages of 18-80.
* Patient population: Males or females who have been previously diagnosed with Neurogenic Orthostatic Hypotension.

Exclusion Criteria:

Patient population:

1. Medical therapies or medications which could interfere with testing of autonomic function.
2. Clinically significant heart disease.
3. Presence of unrelated nerve damage in the peripheral nervous system.
4. Pregnant or breast feeding females.
5. The presence of failure of other organ systems or systemic illness that can affect autonomic function or your ability to cooperate. These include dementia, heart failure, kidney or liver disease, severe anemia, alcoholism, any new and abnormal cell growth identified as malignant, hypothyroidism, surgical procedures where the nerves of the sympathetic nervous system have been cut, or cerebrovascular disease.

Exclusion criteria for monitoring the effects of melatonin

1. All the above PLUS No lying/night time hypertension as determined by 24-hour blood pressure monitoring

Exclusion criteria for healthy controls:

1. Presence of ANY autonomic dysfunction
2. Medical therapies or medications which could interfere with testing of autonomic function.
3. Clinically significant heart disease.
4. Presence of ANY nerve damage in the peripheral nervous system.
5. Pregnant or breast feeding females.
6. The presence of failure of other organ systems or systemic illness that can affect autonomic function or your ability to cooperate. These include dementia, heart failure, kidney or liver disease, severe anemia, alcoholism, any new and abnormal cell growth identified as malignant, hypothyroidism, surgical procedures where the nerves of the sympathetic nervous system have been cut, or cerebrovascular disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Investigation into the integrity of post-ganglionic sympathetic nerves in idiopathic NOH | Sympathetic markers will be assessed during and immediately following the test. A comparison between healthy participants and NOH patients will be ongoing throughout recruitment and upon completion of study recruitment
  Markers of post-ganglionic sympathetic function will be examined (i.e. sympathetic blood markers, heart rate, blood pressure, sympathetic nerve activity, etc.)
Effects of melatonin on supine hypertension in persons with neurogenic orthostatic hypotension | 4 weeks
  Supine systolic blood pressure
Effects of melatonin on supine hypertension in patients with neurogenic orthostatic hypotension | 4 weeks
  Change in postural (supine-standing) systolic blood pressure

SECONDARY OUTCOMES:
Serum markers of sympathetic activation | Before and during stimulation of sympathetic nervous system
Carotid artery diameter | During stimulation of sympathetic nervous system
Sympathetic nerve activation using microneurography | During stimulation of sympathetic nervous system
Orthostatic symptoms based on standard autonomic symptom questionnaires | 30 minutes before testing
Sleep quality assessment using Epworth Sleepiness Scale | Assessed at pre- and post- melatonin treatment; week 1 and week 5 of melatonin intervention timeframe
Urine and Saliva melatonin levels | Assessed at pre- and post- melatonin treatment; week 1 and week 5 of melatonin intervention timeframe

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bendini C, Angelini A, Salsi F, Finelli ME, Martini E, Neviani F, Mussi C, Neri M. Relation of neurocardiovascular instability to cognitive, emotional and functional domains. Arch Gerontol Geriatr. 2007;44 Suppl 1:69-74. doi: 10.1016/j.archger.2007.01.010. PMID 17317436
- [Background] Buscemi N, Vandermeer B, Hooton N, Pandya R, Tjosvold L, Hartling L, Baker G, Klassen TP, Vohra S. The efficacy and safety of exogenous melatonin for primary sleep disorders. A meta-analysis. J Gen Intern Med. 2005 Dec;20(12):1151-8. doi: 10.1111/j.1525-1497.2005.0243.x. PMID 16423108
- [Background] Cagnacci A, Cannoletta M, Renzi A, Baldassari F, Arangino S, Volpe A. Prolonged melatonin administration decreases nocturnal blood pressure in women. Am J Hypertens. 2005 Dec;18(12 Pt 1):1614-8. doi: 10.1016/j.amjhyper.2005.05.008. PMID 16364834
- [Background] Capsoni S, Viswanathan M, De Oliveira AM, Saavedra JM. Characterization of melatonin receptors and signal transduction system in rat arteries forming the circle of Willis. Endocrinology. 1994 Jul;135(1):373-8. doi: 10.1210/endo.135.1.8013371.
- [Background] Cordeiro RC, Jardim JR, Perracini MR, Ramos LR. Factors associated with functional balance and mobility among elderly diabetic outpatients. Arq Bras Endocrinol Metabol. 2009 Oct;53(7):834-43. doi: 10.1590/s0004-27302009000700007. PMID 19942985
- [Background] Freeman R, Wieling W, Axelrod FB, Benditt DG, Benarroch E, Biaggioni I, Cheshire WP, Chelimsky T, Cortelli P, Gibbons CH, Goldstein DS, Hainsworth R, Hilz MJ, Jacob G, Kaufmann H, Jordan J, Lipsitz LA, Levine BD, Low PA, Mathias C, Raj SR, Robertson D, Sandroni P, Schatz I, Schondorff R, Stewart JM, van Dijk JG. Consensus statement on the definition of orthostatic hypotension, neurally mediated syncope and the postural tachycardia syndrome. Clin Auton Res. 2011 Apr;21(2):69-72. doi: 10.1007/s10286-011-0119-5. No abstract available. PMID 21431947
- [Background] Goldstein DS, Sharabi Y. Neurogenic orthostatic hypotension: a pathophysiological approach. Circulation. 2009 Jan 6;119(1):139-46. doi: 10.1161/CIRCULATIONAHA.108.805887. No abstract available. PMID 19124673
- [Background] Grossman E, Laudon M, Yalcin R, Zengil H, Peleg E, Sharabi Y, Kamari Y, Shen-Orr Z, Zisapel N. Melatonin reduces night blood pressure in patients with nocturnal hypertension. Am J Med. 2006 Oct;119(10):898-902. doi: 10.1016/j.amjmed.2006.02.002. PMID 17000226
- [Background] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Influence of circadian time of hypertension treatment on cardiovascular risk: results of the MAPEC study. Chronobiol Int. 2010 Sep;27(8):1629-51. doi: 10.3109/07420528.2010.510230. PMID 20854139
- [Background] Imrich R, Eldadah BA, Bentho O, Pechnik S, Sharabi Y, Holmes C, Grossman E, Goldstein DS. Functional effects of cardiac sympathetic denervation in neurogenic orthostatic hypotension. Parkinsonism Relat Disord. 2009 Feb;15(2):122-7. doi: 10.1016/j.parkreldis.2008.04.002. Epub 2008 May 29. PMID 18514012
- [Background] Pogan L, Bissonnette P, Parent L, Sauve R. The effects of melatonin on Ca(2+) homeostasis in endothelial cells. J Pineal Res. 2002 Aug;33(1):37-47. doi: 10.1034/j.1600-079x.2002.01890.x. PMID 12121484
- [Background] Ray CA. Melatonin attenuates the sympathetic nerve responses to orthostatic stress in humans. J Physiol. 2003 Sep 15;551(Pt 3):1043-8. doi: 10.1113/jphysiol.2003.043182. Epub 2003 Jul 17. PMID 12869610
- [Background] Rich-Edwards JW, Manson JE, Hennekens CH, Buring JE. The primary prevention of coronary heart disease in women. N Engl J Med. 1995 Jun 29;332(26):1758-66. doi: 10.1056/NEJM199506293322607. No abstract available. PMID 7760894
- [Background] Robertson D, Robertson RM. Causes of chronic orthostatic hypotension. Arch Intern Med. 1994 Jul 25;154(14):1620-4. PMID 8031210
- [Background] Rose KM, Eigenbrodt ML, Biga RL, Couper DJ, Light KC, Sharrett AR, Heiss G. Orthostatic hypotension predicts mortality in middle-aged adults: the Atherosclerosis Risk In Communities (ARIC) Study. Circulation. 2006 Aug 15;114(7):630-6. doi: 10.1161/CIRCULATIONAHA.105.598722. Epub 2006 Aug 7. PMID 16894039
- [Background] Satake N, Oe H, Shibata S. Vasorelaxing action of melatonin in rat isolated aorta; possible endothelium dependent relaxation. Gen Pharmacol. 1991;22(6):1127-33. doi: 10.1016/0306-3623(91)90589-x. PMID 1667303
- [Background] Scheer FA, Van Montfrans GA, van Someren EJ, Mairuhu G, Buijs RM. Daily nighttime melatonin reduces blood pressure in male patients with essential hypertension. Hypertension. 2004 Feb;43(2):192-7. doi: 10.1161/01.HYP.0000113293.15186.3b. Epub 2004 Jan 19. PMID 14732734
- [Background] Senard JM, Rascol O, Durrieu G, Tran MA, Berlan M, Rascol A, Montastruc JL. Effects of yohimbine on plasma catecholamine levels in orthostatic hypotension related to Parkinson disease or multiple system atrophy. Clin Neuropharmacol. 1993 Feb;16(1):70-6. doi: 10.1097/00002826-199302000-00008. PMID 8422659
- [Background] Shannon JR, Jordan J, Diedrich A, Pohar B, Black BK, Robertson D, Biaggioni I. Sympathetically mediated hypertension in autonomic failure. Circulation. 2000 Jun 13;101(23):2710-5. doi: 10.1161/01.cir.101.23.2710. PMID 10851208
- [Background] Sharabi Y, Eldadah B, Li ST, Dendi R, Pechnik S, Holmes C, Goldstein DS. Neuropharmacologic distinction of neurogenic orthostatic hypotension syndromes. Clin Neuropharmacol. 2006 May-Jun;29(3):97-105. doi: 10.1097/01.WNF.0000220822.80640.0D. PMID 16772807
- [Background] Stankov B, Capsoni S, Lucini V, Fauteck J, Gatti S, Gridelli B, Biella G, Cozzi B, Fraschini F. Autoradiographic localization of putative melatonin receptors in the brains of two Old World primates: Cercopithecus aethiops and Papio ursinus. Neuroscience. 1993 Jan;52(2):459-68. doi: 10.1016/0306-4522(93)90172-c. PMID 8383820
- [Background] Vagaonescu TD, Saadia D, Tuhrim S, Phillips RA, Kaufmann H. Hypertensive cardiovascular damage in patients with primary autonomic failure. Lancet. 2000 Feb 26;355(9205):725-6. doi: 10.1016/S0140-6736(99)05320-9. PMID 10703810
- [Background] Weekley LB. Effects of melatonin on isolated pulmonary artery and vein: role of the vascular endothelium. Pulm Pharmacol. 1993 Jun;6(2):149-54. doi: 10.1006/pulp.1993.1019. PMID 8358182
- [Background] Cunnane SC, Manku MS, Oka M, Horrobin DF. Enhanced vascular reactivity to various vasoconstrictor agents following pinealectomy in the rat: role of melatonin. Can J Physiol Pharmacol. 1980 Mar;58(3):287-93. doi: 10.1139/y80-049. PMID 7378930
- [Background] Zanoboni A, Forni A, Zanoboni-Muciaccia W, Zanussi C. Effect of pinealectomy on arterial blood pressure and food and water intake in the rat. J Endocrinol Invest. 1978 Apr;1(2):125-30. doi: 10.1007/BF03350359. PMID 755848
- [Background] Zanoboni A, Zanoboni-Muciaccia W. Experimental hypertension in pinealectomized rats. Life Sci. 1967 Nov 1;6(21):2327-31. doi: 10.1016/0024-3205(67)90043-4. No abstract available. PMID 6060280
- [Background] Holmes SW, Sugden D. Proceedings: The effect of melatonin on pinealectomy-induced hypertension in the rat. Br J Pharmacol. 1976 Mar;56(3):360P-361P. No abstract available. PMID 1260192
- [Background] Brown GM, Bar-Or A, Grossi D, Kashur S, Johannson E, Yie SM. Urinary 6-sulphatoxymelatonin, an index of pineal function in the rat. J Pineal Res. 1991 Apr;10(3):141-7. doi: 10.1111/j.1600-079x.1991.tb00831.x. PMID 1880710
- [Background] Briaud SA, Zhang BL, Sannajust F. Continuous light exposure and sympathectomy suppress circadian rhythm of blood pressure in rats. J Cardiovasc Pharmacol Ther. 2004 Jun;9(2):97-105. doi: 10.1177/107424840400900205. PMID 15309246